CLINICAL TRIAL: NCT05003271
Title: Pulmonary Rehabilitation Post-COVID-19: a Pilot Study
Brief Title: Pulmonary Rehabilitation Post-COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Health Sciences Centre Foundation, Manitoba (Other); Health Sciences Centre, Winnipeg, Manitoba (Other)
Responsible Party: Principal Investigator, Diana C Sanchez-Ramirez, PhD, Assistant professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS25183(B2021:101)
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: Long COVID-19; Persistent respiratory symptoms
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Two groups pre-post assessment (pilot/feasibility study)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Small group zoom meeting (Experimental): Group one: participants were asked to follow the exercise program with a small group of peers (2 groups/6 participants each) in a Zoom meeting 3 times a week/45 min each (including 5 min before and 10 min after the meeting for free talk-chat between the participants; e.g., questions, perceptions, etc.).
  Interventions: Other: Exercise program (virtual/remote)
- YouTube pre-recorded video (Experimental): Group two: participants were asked to follow the exercise program 3 times a week/30 min each while watching a pre-recorded YouTube video.
  Interventions: Other: Exercise program (virtual/remote)

INTERVENTIONS:
Other: Exercise program (virtual/remote) — Intervention (8 weeks): using the participants' initial assessment and personal characteristics, the therapist will provide personalized recommendations (e.g. maximum heart rate, minimum SpO2), explain the educational materials, and instruct patients on safety precautions.

SUMMARY:
The main objective of this pilot study was to evaluate the feasibility, safety, and satisfaction of a remote interdisciplinary PR program delivered using two exercise approaches (video conference and self-directed) on the recovery of long-term post-COVD-19 outcomes. The specific aims were i) to evaluate the effect of each of the approaches on patients': 1) lung capacity, 2) dyspnea and fatigue, 3) exercise capacity, 4) physical function, 5) participation, and 5) HRQoL.

DETAILED DESCRIPTION:
This pilot study used a two-arm randomized pre- and post-trial design to evaluate the feasibility, safety, and satisfaction of a remote interdisciplinary PR program, delivered using two exercise approaches (video conference and self-directed), on the recovery of long-term post-COVD-19 outcomes (≥ 3 months after infection). Group one (video conference): participants were asked to follow the exercise program with a small group of peers (2 groups/6 participants each) in a Zoom meeting 3 times a week/45 min each (including 5 min before and 10 min after the meeting for free talk-chat between the participants; e.g. questions and perceptions). The therapist organized and led the Zoom meetings to resolve general questions (e.g. equipment, platforms, etc.). Group two: participants were asked to follow the exercise program 3 times a week/30 min each while watching a pre-recorded video created by the research team and uploaded on YouTube. Patients were asked to wear the finger pulse oximeter at all times while exercising, so that they could control their pace while avoiding exceeding target values (HR and SpO2). They were also asked to record their HR and SpO2 values before and after participation in every session of the exercise program in a diary. All participants from both groups could contact the therapist at any time during the study if they had questions or concerns. They also received a follow-up phone call once a week from the therapist.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID-19 ≥ 3 months after infection.
* Mild to severe persistent respiratory symptoms
* Access to a smart phone, tablet or computer, and home internet

Exclusion Criteria:

* History of neurological disease or mental illness
* Inability to ambulate independently without supervision
* Inability to complete basic tasks on a smart phone or tablet
* Did not return calls after the initial contact

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of the program | 8 weeks (end of the study)
  This was determined according to the following criteria: (1) 70% of participants completed the PR program, (2) data on primary outcomes collected in ≥ 70% of participants after the PR program, and (3) < 10% of adverse events related to the intervention.
Recruitment rate | 8 weeks (beginning of the study)
  Calculated as percentage of potentially eligible participants that were recruited.
Intervention completion rate | 8 weeks
  Calculated as the percentage of sessions attended by participants. The number of sessions in the vide conference group was recorded by the therapist who attended Zoom meeting, whereas those in the self-directed group were asked to record the number of sessions in the diary.
Dropout rate | 8 weeks
  Calculated as the proportion of individuals who ceased participation after randomization and before completing 80% of sessions due to adverse events or personal preferences.
Patient safety | 8 weeks
  Represented as the incidence of adverse events caused by the interventions.
Patient satisfaction with the program | after 8 weeks (end of the study)
  Participants will complete a short summary with questions regarding their satisfaction with the study

SECONDARY OUTCOMES:
Change in lung capacity | 8 weeks
  It was assessed using a SpiroBank Smart F/V multi parameter spirometer (MIR) at pre-post intervention and once a week in between to monitor changes. This portable spirometer, which is MDSAP approved and complaint with ATS/ERS guidelines, connects automatically via Bluetooth to an iOS & Android compatible App (MIR Spirobank). It provides real time feedback through messages and animation on smartphone, to improve personal compliance during the test. The app can generate test results PDF printout with information regarding 19 parameters of lung capacity. The following main variables were used: forced vital capacity, forced expiratory volume in the first second, ratio between forced expiratory volume in the first second and forced vital capacity, and peak expiratory flow.
Change in dyspnea | 8 weeks
  Modified Borg Scale (0 "best" to 10 "worse") was used to assess dyspnea.
Changes in fatigue severity assessed with the Fatigue Severity Scale | 8 weeks
  The Fatigue Severity Scale (0 -7 "higher worse") was used to measure the severity of fatigue. Overall fatigue severity was assessed using the visual analog scale included in the Fatigue Severity Scale (0 "worst" - 10"normal").
Changes in fatigue assesses with the DePaul Symptom Questionnaire short-form | 8 weeks
  The DePaul Symptom Questionnaire short-form assessed the frequency and severity of 14 symptoms (0 - 100, "higher is worst") related to fatigue at rest, post-exertional fatigue, pain, and neurocognitive, autonomic/neuroendrocrine, and immune systems.
Change in sit-to-stand capacity | 8 weeks
  Sit-to-stand capacity was used as a measure of exercise capacity. It was assessed using the one-minute sit-to-stand test (number of times the persons can complete the task in one minute).
Change in post-exercise saturation | 8 weeks
  SpO2 will be measured using a digital fingertip pulse oximeter (LOOKEE®, New York, USA) before-after the one- minute sit-to-stand test.
Change in HRQoL | 8 weeks
  Assessed using the EQ-5D-5L scale (https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/)(mobility, self-care, usual activities, pain/discomfort and anxiety/depression). General health was assessed using a visual analog scale (EQVAS): 0 (worst imaginable health state) and 100 (best imaginable health state today).
Change in activities participation | 8 weeks
  Assessed using the Canadian Occupational Performance Measure (COPM) which focuses on occupational performance in all areas of life, including self-care, leisure, and productivity.
Feasibility of collecting data using wearable technology | 1 week
  A subgroup of participants were asked to use a wrist-worn smartwatch and waist-worn accelerometer (non-dominant hip) for seven days.

CONTACTS AND LOCATIONS:
Overall Officials: Diana C Sanchez-Ramirez, PhD, Principal Investigator — University of Manitoba
Locations (1):
- U of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sarmento A, Adodo R, Hodges G, Webber SC, Sanchez-Ramirez DC. Virtual pulmonary rehabilitation approaches in patients with post COVID syndrome: a pilot study. BMC Pulm Med. 2024 Mar 18;24(1):139. doi: 10.1186/s12890-024-02965-3. PMID 38500051